CLINICAL TRIAL: NCT06088290
Title: Randomized, Controlled, Open-label, Phase III Study of Lurbinectedin in Combination With Doxorubicin Versus Doxorubicin Alone as First-line Treatment in Patients With Metastatic Leiomyosarcoma
Brief Title: Study of Lurbinectedin in Combination With Doxorubicin Versus Doxorubicin Alone as First-line Treatment in Participants With Metastatic Leiomyosarcoma (SaLuDo)
Acronym: SaLuDo
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-C-010-22; 2022-502975-45 (EudraCT Number)
Record Dates: First submitted 2023-09-28; First posted 2023-10-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Leiomyosarcoma
Keywords: Leiomyosarcoma; Oncology
MeSH Terms: conditions — Leiomyosarcoma; Neoplasms | interventions — PM 01183; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Doxorubicin (Dose A) + Lurbinectedin (Dose B) (Experimental): Participants will receive doxorubicin and lurbinectedin intravenously (IV) every three weeks (q3wk) on Day 1 of each treatment cycle (treatment cycle = three weeks).
  Interventions: Drug: Lurbinectedin; Drug: Doxorubicin
- Doxorubicin (Dose C) + Lurbinectedin (Dose D) (Experimental): Participants will receive doxorubicin IV q3wk on Day 1 of each treatment cycle (treatment cycle = three weeks).
  Interventions: Drug: Lurbinectedin; Drug: Doxorubicin
- Doxorubicin (Active Comparator): Participants will receive doxorubicin IV q3wk on Day 1 of each treatment cycle (treatment cycle = three weeks).
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Lurbinectedin — IV Infusion
  Arms: Doxorubicin (Dose A) + Lurbinectedin (Dose B); Doxorubicin (Dose C) + Lurbinectedin (Dose D)
Drug: Doxorubicin — Short IV push or bolus (according to label)

SUMMARY:
The primary objective of this phase III study is to evaluate whether the combination of lurbinectedin plus doxorubicin given as first line treatment for metastatic leiomyosarcoma (LMS) prolongs the progression-free survival (PFS) by Independent Review Committee (IRC) when compared to doxorubicin administered as a single agent.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed and dated written informed consent of the participants obtained before any study-specific procedure.
2. Age ≥ 18 years.
3. Histologically confirmed diagnosis of metastatic LMS, in participants not candidates for curative resection.
4. Radiologically measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
5. No previous systemic therapy for metastatic disease (i.e., first-line setting) and no previous anthracyclines. Note: prior chemotherapy (without anthracycline) in the context of adjuvant or neoadjuvant therapy is allowed. Prior line/s of hormone therapy in the adjuvant/metastatic setting are also allowed.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
7. Adequate hematological, renal, metabolic and hepatic function:

   1. Hemoglobin ≥ 9.0 g/dL (participants may have received prior red blood cell [Red Blood Cell] transfusion); absolute neutrophil count (ANC) ≥ 2.0 x 10^9/L, and platelet count

      ≥ 100 x 10^9/L.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x upper limit of normal (ULN).
   3. Total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN if total bilirubin is > ULN.
   4. Albumin ≥ 3.0 g/dL.
   5. Calculated creatinine clearance (CrCL) ≥ 30 mL/min (using Cockcroft and Gault's formula).
   6. Left ventricular ejection fraction (LVEF) > 50% assessed by multiple-gated acquisition scan (MUGA) or echocardiography (ECHO) or cardiac magnetic resonance imaging (MRI).
8. Wash-out periods:

   1. At least three weeks since last prior systemic treatment.
   2. At least three weeks since last prior major surgery and one week since last prior minor surgery (port placement is excluded from this wash-out period).
   3. At least two weeks since last prior radiotherapy.
9. Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure up to seven months after treatment discontinuation. Fertile male participants with WOCBP partners should use condoms during treatment and for four months following the last investigational medicinal product (IMP) dose.

Exclusion Criteria:

1. Prior treatment with anthracyclines, lurbinectedin or trabectedin.
2. Known low grade leiomyosarcoma (i.e., grade I).
3. Known hypersensitivity to any of the components of the IV formulation of lurbinectedin or doxorubicin.
4. Concomitant diseases/conditions:

   1. History of cardiac disease: myocardial infarction or angina within the year prior to enrollment; severe vascular disease; or symptomatic arrhythmia despite ongoing treatment.
   2. Participants with any immunodeficiency, including those known to be infected by human immunodeficiency virus (HIV).
   3. Known chronic active hepatitis or cirrhosis. For Hepatitis B, this includes positive tests for both Hepatitis B surface antigen and quantitative Hepatitis B polymerase chain reaction (PCR). For Hepatitis C, this includes positive tests for both Hepatitis C antibody and quantitative Hepatitis C PCR.
   4. Active uncontrolled infection.
   5. Any other major illness that (including severe cardiovascular disease) or risk factors that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
5. Use of strong inducers of CYP3A4 activity within two weeks prior to the first infusion of lurbinectedin.
6. Prior irradiation of a RECIST v.1.1 target lesion if only one target lesion is available, unless progression of the lesion has been confirmed.
7. Known myopathy (history of resolved steroid-induced myopathy is allowed).
8. History of malignancies other than LMS within three years prior to enrollment, except for malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, non-muscle-invasive urothelial carcinomas, ductal carcinoma in situ, or stage I uterine cancer. Prior malignancies should have received curative treatment and should remain in remission. The Investigator should ensure, based on histology or clinical information, that the current metastatic sites are leiomyosarcoma and not recurrence of the original malignancy.
9. Limitation of the participant's ability to comply with the treatment or to follow-up the protocol.
10. Women who are pregnant or breast feeding and fertile participants (men and women) who are not using a highly effective method of contraception.
11. Participants in whom rapid tumor shrinkage is needed (e.g., when a tumor is close to a critical structure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
PFS by IRC | Up to approximately 41 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 66 months
PFS by Investigator's Assessment (IA) | Up to approximately 41 months
Overall Response Rate (ORR) by IRC and IA | Up to approximately 66 months
Duration of Response (DoR) by IRC and IA | Up to approximately 66 months
Clinical Benefit Rate (CBR) by IRC and IA | Up to approximately 66 months
PFS on Next-line Therapy (PFS2) by IA | Up to approximately 41 months
Number of Participants Experiencing Adverse Events (AE) | Up to approximately 66 months
Number of Participants Experiencing Serious Adverse Events (SAE) | Up to approximately 66 months
Change in Quality of Life by European Organization for Research and Treatment of Cancer (EORTC) 30-item Quality of Life Questionnaire (QLQ-C30) | Up to approximately 41 months
Clearance of Lurbinectedin and Doxorubicin in the Plasma | Cycle 1 Day 1, and Day 5 (One cycle = 3 weeks)
Volume of Distribution of Lurbinectedin and Doxorubicin in the Plasma | Cycle 1 Day 1, and Day 5 (One cycle = 3 weeks)
Number of Participants With Presence or Absence of Mutation per Molecular Biomarker Associated With Response and/or Resistance to Treatment | Up to approximately 41 months
Expression Levels of Molecular Biomarkers Associated with Response and/or Resistance to Treatment | Up to approximately 41 months

CONTACTS AND LOCATIONS:
Locations (94):
- United States (22):
  - Mayo Clinic Hospital - Phoenix, Phoenix, Arizona
  - Precision NextGen Oncology & Research Center, Beverly Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarcoma Oncology Center, Los Angeles, California
  - Stanford University (Leland Stanford Junior University), Palo Alto, California
  - University of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center - New York, New York, New York
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center - Seattle Cancer Care Alliance (SCCA) Location, Seattle, Washington
- Austria (4):
  - Universitaetsklinikum Graz - Universitätsklinik für Innere Medizin, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Medizinische Universität Wien, Vienna
- Belgium (4):
  - Universitair Ziekenhuis Bruseel, Jette, Brussels Capital
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- France (13):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional et Universitaire de Besançon - Hôpital Jean-Minjoz, Besançon, Doubs
  - Institut de Cancérologie de l'Ouest - Angers, Angers, Pays de la Loire Region
  - Centre Antoine Lacassagne, Nice, Provence-Alpes-Côte d'Azur Region
  - Institut Bergonié, Bordeaux
  - Centre de Lutte contre le Cancer - Centre Oscar Lambret, Lille
  - Centre Hospitalier Universitaire Dupuytren 1, Limoges
  - Hôspital de la Timone, Marseille
  - Institut Curie, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest - Saint-Herblain - Site René Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif
- Germany (8):
  - LMU Klinikum - Campus Großhadern, München, Bavaria
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mannheim, Manheim
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
- Italy (12):
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Istituto Clinico Humanitas, Rozzano, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Naples
  - Centro di Riferimento Oncologico, Aviano
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico Sant Orsola-Malpighi, Bologna
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Università Campus Bio-Medico di Roma, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino
- Netherlands (2):
  - Het Nederlands Kanker Instituut, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum (LUMC), Leiden, South Holland
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Szpitale Pomorskie Spółka Z Ograniczoną Odpowiedzialnością, Gdynia, Pomeranian Voivodeship
- Portugal (4):
  - Instituto Portugues De Oncologia De Lisboa Francisco Gentil, Lisbon, Lisbon District
  - Unidade Local de Saúde de Coimbra, Coimbra
  - Unidade Local de Saúde de Santo António, E.P.E - Hospital Geral de Santo António, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, Porto
- Spain (14):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - START Madrid - CIOCC - HM Sanchinarro, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
- United Kingdom (7):
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cote GM, Chawla SP, Demetri G, Kasper B, Jones RL, Broto JM, Wooley J, Weiss MC, Tafuto S, Badalamenti G, Carrasco I, Peinado P, Blay JY, Boggio G, Fernandez C, Nieto A, Kahatt C, Alfaro V, Le Cesne A. SaLudo: a randomized phase IIb/III study of lurbinectedin plus doxorubicin as first-line treatment in leiomyosarcoma. Future Oncol. 2025 Apr;21(8):943-951. doi: 10.1080/14796694.2025.2463798. Epub 2025 Feb 11. PMID 39932221